CLINICAL TRIAL: NCT02328287
Title: A Pilot Phase 2a, Multicentre, Open, Proof-of-concept Study on the Safety and the Efficacy of Allogeneic Osteoblastic Cells (ALLOB®) Implantation in Rescue Interbody Fusion
Brief Title: Study on Allogeneic Osteoblastic Cells Implantation in Rescue Interbody Fusion
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bone Therapeutics S.A (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLOB-RIF1
Record Dates: First submitted 2014-12-23; First posted 2014-12-31 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Failed Lumbar Fusion
Keywords: Spinal Fusion; Revision Surgery; Pseudarthrosis; Cell Therapy; Bone Graft
MeSH Terms: conditions — Pseudarthrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALLOB® Implantation (Experimental)
  Interventions: Drug: ALLOB®

INTERVENTIONS:
Drug: ALLOB® — Each patient will undergo a single administration of ALLOB® into the failed fusion lumbar level under anesthesia.

SUMMARY:
Failed fusion and failure to relieve back pain following spinal fusion are still frequent, irrespective of the type of procedures or grafts used by the surgeon. Moreover, revision surgeries are unfortunately associated with higher procedure-related complication rates, technical difficulties, longer operative time, and quite disappointing and unreliable success rates for both fusion and clinical results.

The present Phase 2a study aims at demonstrating the safety and efficacy of ALLOB®, a proprietary population of allogeneic osteoblastic cells, in rescue interbody fusion.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide a written, dated, and signed informed consent prior to any study related procedure, and to understand and comply with study requirements
* Failed lumbar fusion of 15 months minimum requiring a revision surgery at one or two levels between L1 and S1

Exclusion Criteria:

* More than two failed interbody fusions at the involved lumbar level(s)
* Instrumentation failure requiring revision surgery
* Local active or latent infection at the involved lumbar level(s)
* Positive serology for hepatitis B, hepatitis C, HIV
* Current or past medical disease that could interfere with the evaluation of the safety and efficacy, as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Lumbar fusion progression as assessed by CT scan | 12 months
Functional Disability using Oswestry Disability Index | 12 months
Potential occurrence of any AE or SAE, related to the product or to the procedure, using patient open non-directive questionnaire, physical examination and laboratory measurements | 12 months

SECONDARY OUTCOMES:
Pain using a Visual Analogue Scale | 12 months
Global Disease Evaluation using a Visual Analogue Scale | 12 months
Functional Disability using Oswestry Disability Index | 12 months
Lumbar fusion progression as assessed by CT scan | 12 months
Percentage of patients having a rescue surgery | 12 months
Potential occurrence of any AE or SAE, related to the product or to the procedure, using patient open non-directive questionnaire, physical examination and laboratory measurements | 36 months

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Investigating site BE01, Anderlecht
  - Investigating site BE02, Charleroi
  - Investigating site BE04, Genk